CLINICAL TRIAL: NCT00628511
Title: A Validation Study of A New Diagnostic Device for Screening of Obstructive Sleep Apnea in High Risk Patient Population
Brief Title: Validation of Portable Monitoring Device for Diagnosing Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: To K W, The Hospital Authority
Other Study IDs: 6902256
Record Dates: First submitted 2008-02-06; First posted 2008-03-05 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2008-02

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observation
  Interventions: Device: ARES (Apnea Risk Evaluation System)

INTERVENTIONS:
Device: ARES (Apnea Risk Evaluation System) — application of portable monitoring device with PSG

SUMMARY:
portable monitoring device could diagnose sleep apnea in high risk patients.

DETAILED DESCRIPTION:
This is a pilot study of another larger cohort investigating different algorithms in managing patients suspected of sleep apnea using portable monitoring device.

Portable monitoring device is applied simultaneously with PSG to compare it's accuracy and validity.

ELIGIBILITY:
Inclusion Criteria:

* patients suspected of sleep apnea

Exclusion Criteria:

* patient refuse to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients suspected of sleep apnea
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
validity of portable monitoring device | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: To K Wang, MBCHB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese Univerisity of Hong Kong, Hong Kong, China